CLINICAL TRIAL: NCT01614600
Title: Clinical Evaluation of a Daily Disposable Contact Lens in Symptomatic Weekly/Monthly Lens Wearers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A00849
Record Dates: First submitted 2012-06-06; First posted 2012-06-08 (Estimated); Results first posted 2013-12-04 (Estimated); Last update posted 2013-12-04 (Estimated); Status verified 2013-09

CONDITIONS: Dry Eye Syndrome; Myopia
Keywords: contact lens; dry eye syndrome; symptomatic; daily disposable; myopia
MeSH Terms: conditions — Dry Eye Syndromes; Myopia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- DAILIES® AquaComfort Plus® (Experimental): Nelfilcon A contact lenses worn bilaterally on a daily wear, daily disposable basis for 2 weeks
  Interventions: Device: Nelfilcon A contact lenses

INTERVENTIONS:
Device: Nelfilcon A contact lenses — Commercially marketed hydrogel contact lenses for daily wear, daily disposable use
  Other Names: DAILIES® AquaComfort Plus®

SUMMARY:
The purpose of this study was to evaluate the reduction of contact lens-related dryness symptoms when symptomatic weekly/monthly contact lens wearers were switched to DAILIES® AquaComfort Plus® lenses for a two-week period using composite scores on the Contact Lens Dry Eye Questionnaire (CLDEQ).

ELIGIBILITY:
Inclusion Criteria:

* Currently wearing weekly/monthly, silicone hydrogel or traditional hydrogel soft contact lenses at least 8 hours per day and 5 days a week during the past 6 months.
* Identified as symptomatic using a baseline screening questionnaire.
* Requires vision correction in both eyes with a contact lens prescription as follows: sphere powers between -0.50 and -10.00 diopter (D) and cylinder powers </= 0.75D and no ADD correction.
* Able to achieve visual acuity (VA) of at least 6/7.5 in each eye with study lenses in the available parameters.
* Willing to wear study lenses for at least 8 hours/day and at least 5 days/week and discard the lenses at the end of the day and replace lenses every day with a new fresh pair.
* Willing and able to follow instructions and maintain the appointment schedule.
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Neophytes and current wearers of daily disposable contact lenses.
* Requires monovision correction.
* Any systemic or ocular disease or disorder (refractive disorder allowed) complicating factors or structural abnormality that would negatively affect the conduct or outcome of the study.
* A history of ocular surgery/trauma within the last 6 months.
* Unwilling to discontinue mechanical eyelid therapy or eyelid scrubs within 14 days of enrollment and continuing during the study.
* Participation in any other ophthalmic drug or device clinical trial within 30 days of enrollment.
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2012-06; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jami Kern, MBA, PhD, Study Director — Alcon Research

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from 8 study centers located in the United States.
Pre-assignment Details: Of the 91 participants enrolled, 3 were exited as screen failures prior to dispensing of the study product. This reporting group includes all enrolled and dispensed participants.
Period: Overall Study
Arm/Group | DAILIES® AquaComfort Plus®
Started | 88
Completed | 84
Not Completed | 4
Not completed — Unacceptable fit | 1
Not completed — Discomfort | 1
Not completed — Unable to remove lens at the end of day | 1
Not completed — Protocol deviation | 1

BASELINE CHARACTERISTICS:
Population: This reporting group includes all enrolled and dispensed participants.
Arm/Group | DAILIES® AquaComfort Plus®
Number analyzed (Participants) | 88
Age Continuous [Mean (Standard Deviation); unit: years] | 32.2 (9.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 66
  Male | 22
Region of Enrollment [Number; unit: participants]
  United States | 88

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Contact Lens-Related Dryness Symptoms at Week 1 and Week 2
Description: Contact lens symptoms were evaluated using the Contact Lens Dry Eye Questionnaire (CLDEQ). Subjects rated 8 common contact lens-related ocular surface dryness symptoms at Baseline, Week 1, and Week 2 using a 5-point scale (1=never or not at all intense, 5=constantly or very intense). A scoring algorithm was used to calculate a composite score for each visit for all symptoms (-6.5 to 10). A higher composite score would indicate more contact lens related dry eye and a lower score, less contact lens related dry eye.
Time Frame: Baseline, Week 1, Week 2
Population: Per Protocol: All enrolled and dispensed participants, minus any major protocol deviators as determined by masked review.
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | DAILIES® AquaComfort Plus®
Number analyzed (Participants) | 74
Units on a scale
  Change from Baseline at Week 1 | -0.09 (1.24)
  Change from Baseline at Week 2 | -0.29 (1.06)

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study (3 months).
Description: This reporting group includes all enrolled and dispensed participants.
Arm/Group | DAILIES® AquaComfort Plus®
Serious Adverse Events (participants affected / at risk) | 0/88
Other Adverse Events (participants affected / at risk) | 0/88

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor reserves the right of prior review of any publication or presentation of information related to the study.